CLINICAL TRIAL: NCT05422261
Title: The Relationship Between Parents' Fatigue and Quality of Life, and the Quality of Life and Participation of Children With Autism Spectrum Disorder
Brief Title: The Relationship Between Parents' Fatigue and Quality of Life
Status: Completed | Type: Observational
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Ozgun Kaya Kara, Assoc. Prof., Akdeniz University
Other Study IDs: 2019/288
Record Dates: First submitted 2022-06-14; First posted 2022-06-16 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; Quality of life; Participation; Depression
MeSH Terms: conditions — Autism Spectrum Disorder; Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental Group: Children with Autism Spectrum Disorder and their parents
- Control Group: Health children and their parents

SUMMARY:
By comparing them to a healthy control group, this study aims to investigate the relationship between the participation of children with autism spectrum disorder (ASD) in home, school, and community environments and their parents' fatigue, depression, and quality of life, as well as the child's quality of life. There is no study that investigators are aware of that looks into the relationship between the fatigue and quality of life of parents of children with ASD and the quality of life and participation of children with ASD. This study hypothesizes that parents of children with ASD experience more fatigue and have a lower health-related quality of life than parents of healthy children.

DETAILED DESCRIPTION:
ASD is a neurodevelopmental disorder characterized by difficulties with social communication, limited and repetitive activities, and sensory sensitivity. The social, emotional, and behavioral issues that children with ASD face are a source of concern for their parents. Mental health issues such as stress, depression, and anxiety are common in these households. According to studies, mothers of children with ASD experience more stress and depression than mothers of children without ASD or mothers of children with other chronic disorders. Another aspect of having an ASD child that has an influence on health is fatigue. In terms of the health of parents of children with ASD, fatigue is often overlooked in study and practice. One of the study was investigated at the fatigue levels of 50 mothers of children with ASD who were between the ages of 2 and 5. Compared to mothers of healthy children, mothers of children with ASD reported higher fatigue, stress, worry, and depressive symptoms.

Participation in daily activities is critical for all children's healthy development, whether or not they have a disability. Participating in activities allows children to express themselves, find purpose, and improve their health. Exclusion and loneliness can arise from a child's inability to participate in normal childhood activities. This circumstance has a number of harmful consequences for the child. According to research, children with ASD participate in their home, school, and community surroundings at a considerably lower rate than their healthy peers, and this difference grows over time.

There is no study in the literature that examines the association between children with ASD's participation in home, school, and community environments, their parents' fatigue level, and the child's quality of life. As a result, the purpose of this research is to look at the relationship between ASD children's participation in home, school, and community settings and their parents' fatigue, depression, and quality of life, as well as the child's quality of life, by comparing them to a healthy control group.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Autism Spectrum Disorder and their parents
* Aged at 2-17 years.
* To be the native language Turkish

Exclusion Criteria:

* Diagnosis of other neurologic disorder such as epilepsy, diabetes, congenital heart disease, brain trauma
* Not to accept to attend the study

Inclusion criteria for control group:

1. Ages at 2-18 years.
2. Not having any psychiatric or neurological diagnosis.
3. To be the native language Turkish.

Exclusion criteria for control group:

1. Not agree to participate the study.
2. To have received medical treatment for any neuropsychiatric disorder.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with diagnosed Autism Spectrum Disorder and their health peers and their families
Sampling Method: Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-05-16 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of fatigue | baseline
  Fatigue Impact Scale is a multidimensional scale that measures the physical, cognitive, and social effects of fatigue. It consists of 40 items divided into 10 cognitive, 10 physical, and 20 social subscales. Each question is scored on a five-point Likert scale from 0 (no problem) to 4 (extreme problem). The maximum score is 160.
Evaluation of fatigue severity | Baseline
  The Fatigue Severity Scale is one of the most commonly used scales to assess fatigue. There are nine questions. Each question is scored on a seven-point Likert scale from one to seven. The mean of nine questions is the scale value.The minimum score is 1 and maximum score is 7. Higher scores indicate more severe fatigue. Although there is no recommendation, it is usually considered that fatigue severity above 4 points is significant.
Evaluation of Quality of Life of children | Baseline
  Quality of Life in Autism Questionnaire-Parent Version is divided into 2 parts (A and B). Part A consists of 28 questions that assess parents' perceptions of their own life quality. Each question is scored on a five-point Likert scale from one (not at all) to five (very much). Part B assesses parents' perceptions of the severity of their child's autism-related difficulties with 20 questions. Each question is scored on a five-point Likert scale from one (not much of a problem for me) to five (very much of a problem for me). Higher scores indicate that a child's autism-related difficulties cause fewer problems for parents. The scale produces a score ranging from minimum 48 to maximum 240 score.

SECONDARY OUTCOMES:
Evaluation of health | Baseline
  Nottingham Health Profile assesses the physical, emotional, and health problems perceived by a person. It consists of 6 different subcategories such as energy, pain, physical mobility, sleep, emotional reactions, and social isolation, with 38 items. Nottingham Health Profile examines the current state of health, and the answers are binary (yes/no).The overall value is calculated by multiplying the intensity of the questions by the positive answer to each one. Minimum score is 0 and maximum score is 100.
Evaluation of depression | Baseline
  Beck Depression Inventory assesses characteristic attitudes and depression symptoms with 21 self-reported items. It takes about 10 minutes to finish the assessment. It is intended for people aged 13 and up. Beck Depression Inventory includes 21 questions. For each question, the lowest score is 0 and the maximum score is 3. The total score of all answers is evaluated as follows 0 to 9 points: "minimal depressive symptoms", 10 to 16 points: "mild depressive symptoms", 17 to 29 points: "moderate depressive symptoms", 20 to 63 points: "severe depressive symptoms".
Evaluation of participation | Baseline
  Participation and Environment- Children and Youth is a parent-reported questionnaire to assess participation and environmental factors in the home, at school, and within community settings. The participation sections included 10 activities in the home setting, five activities in the school setting and 10 in the community setting. For each activity, parents are asked to determine the participation frequency (how frequently has the child participated with eight options: daily to never); participation involvement (how involved the child is while participating in the activity rated on a five-point scale: very involved to minimally involved); and whether change is desired (do the parents want to see change in the child's participation in this type of activity: no or yes, with five different types of change). The minimum score is 0 and the maximum score is 100.

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Results will be presented in the journal

REFERENCES:
- [Result] Battle DE. Diagnostic and Statistical Manual of Mental Disorders (DSM). Codas. 2013;25(2):191-2. doi: 10.1590/s2317-17822013000200017. No abstract available. PMID 24413388
- [Result] Lecavalier L, Leone S, Wiltz J. The impact of behaviour problems on caregiver stress in young people with autism spectrum disorders. J Intellect Disabil Res. 2006 Mar;50(Pt 3):172-83. doi: 10.1111/j.1365-2788.2005.00732.x. PMID 16430729
- [Result] Cohrs AC, Leslie DL. Depression in Parents of Children Diagnosed with Autism Spectrum Disorder: A Claims-Based Analysis. J Autism Dev Disord. 2017 May;47(5):1416-1422. doi: 10.1007/s10803-017-3063-y. PMID 28214978
- [Result] Hayes SA, Watson SL. The impact of parenting stress: a meta-analysis of studies comparing the experience of parenting stress in parents of children with and without autism spectrum disorder. J Autism Dev Disord. 2013 Mar;43(3):629-42. doi: 10.1007/s10803-012-1604-y. PMID 22790429
- [Result] Higgins DJ, Bailey SR, Pearce JC. Factors associated with functioning style and coping strategies of families with a child with an autism spectrum disorder. Autism. 2005 May;9(2):125-37. doi: 10.1177/1362361305051403. PMID 15857858
- [Result] Giallo R, Wood CE, Jellett R, Porter R. Fatigue, wellbeing and parental self-efficacy in mothers of children with an autism spectrum disorder. Autism. 2013 Jul;17(4):465-80. doi: 10.1177/1362361311416830. Epub 2011 Jul 25. PMID 21788255
- [Result] Seymour M, Wood C, Giallo R, Jellett R. Fatigue, stress and coping in mothers of children with an autism spectrum disorder. J Autism Dev Disord. 2013 Jul;43(7):1547-54. doi: 10.1007/s10803-012-1701-y. PMID 23124359
- [Result] King G, Law M, King S, Rosenbaum P, Kertoy MK, Young NL. A conceptual model of the factors affecting the recreation and leisure participation of children with disabilities. Phys Occup Ther Pediatr. 2003;23(1):63-90. PMID 12703385
- [Result] Simpson K, Adams D, Bruck S, Keen D. Investigating the participation of children on the autism spectrum across home, school, and community: A longitudinal study. Child Care Health Dev. 2019 Sep;45(5):681-687. doi: 10.1111/cch.12679. Epub 2019 May 20. PMID 31041826
- [Result] Egilson ST, Jakobsdottir G, Olafsdottir LB. Parent perspectives on home participation of high-functioning children with autism spectrum disorder compared with a matched group of children without autism spectrum disorder. Autism. 2018 Jul;22(5):560-570. doi: 10.1177/1362361316685555. Epub 2017 Apr 21. PMID 28429605
- [Result] Taheri A, Perry A, Minnes P. Examining the social participation of children and adolescents with Intellectual Disabilities and Autism Spectrum Disorder in relation to peers. J Intellect Disabil Res. 2016 May;60(5):435-43. doi: 10.1111/jir.12289. PMID 27120987